CLINICAL TRIAL: NCT02622022
Title: Palliation of Dyspnea With Morphine in Patients With Interstitial Lung Disease
Acronym: MORPHILD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Skanderbog Apotek (Other)
Responsible Party: Principal Investigator, Charlotte Andersen, MD, PhD, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-002533-22
Record Dates: First submitted 2015-12-02; First posted 2015-12-04 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Interstitial Lung Disease; Dyspnea; Morphine
Keywords: randomised; placebo controlled; clinical trial
MeSH Terms: conditions — Lung Diseases, Interstitial; Dyspnea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Morphine (Active Comparator): 18 patients treated with oral morphine hydrochloride linctus 5 mg 4 four times daily and as needed up to 4 times daily
  Interventions: Drug: Morphine hydrochloride
- Placebo (Placebo Comparator): 18 patients treated with oral linctus corresponding to 5 mg morphine hydrochloride, four times daily and as needed up to 4 times daily
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Morphine hydrochloride
  Other Names: Placebo
  Arms: Morphine
Other: Placebo
  Arms: Placebo

SUMMARY:
36 patients with interstitial lung disease will be randomized to 1 weeks treatment with morphine hydrochloride as oral linctus 5 mg, four times a day, and 5 mg as needed up to 4 times a day, or corresponding doses of placebo.

VAS score for dyspnea will be evaluated after 1 hour and 1 week at follow up. Other questionnaires will also be evaluated (GAD-7, K-BUILD, Leicester score)

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of interstitial lung disease (IPF, NSIP, RA-ILS, Scl-ILS, MCTD-ILS, asbestous, drug induced ILD, unclassified ILD)
* Dyspnea corresponding to Medial Research Councils (MRC) dyspnea score ≥ 3
* Written consent
* Age ≥ 18 years
* Competent
* For fertile women: Negative pregnancy test
* For fertile and sexually active participants: Use of safe anti-conceptionals

Exclusion Criteria:

* Ongoing infection
* Decreased lung function to a degree which makes any form of respiratory depression life threatening
* Treatment with morphine or morphine analogues
* Allergy towards morphine hydrochloride

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-01; Primary Completion 2019-02-06 (Actual); Study Completion 2019-02-06 (Actual)

PRIMARY OUTCOMES:
VAS dyspnea score | 1 week

SECONDARY OUTCOMES:
Oxygen saturation | 1 hour and 1 week
  Peripheral oxygen saturation will be measured after first dose of morphine and placebo as well as after 1 week follow up
K-bild questionnaire | 1 week
  questionnaire regarding interstitial lung specific life quality
GAD-7 questionnaire | 1 week
  VAlidatet score for anxiety and depression
6 min walk test | 1 hour and 1 week
Leicester Score | 1 week
  cough related score

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus C, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kronborg-White S, Andersen CU, Kohberg C, Hilberg O, Bendstrup E. Palliation of chronic breathlessness with morphine in patients with fibrotic interstitial lung disease - a randomised placebo-controlled trial. Respir Res. 2020 Jul 23;21(1):195. doi: 10.1186/s12931-020-01452-7. PMID 32703194